CLINICAL TRIAL: NCT01864239
Title: The Medicines Advice Service: A Randomised Controlled Trial of a Pharmacy-based Telephone Intervention to Support Patients Taking Medication for a Long-term Condition
Brief Title: The Medicines Advice Service Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Pharmacy2U (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12/0326
Record Dates: First submitted 2013-04-29; First posted 2013-05-29 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes; Hyperlipidemias
Keywords: Adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient-centred tailored intervention (Experimental): Medicines Advice Service
  Interventions: Other: Medicines Advice Service
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Medicines Advice Service — The intervention consists of:
  1. Telephone consultations with a pharmacist
  2. Follow-up tailored written information
  3. A medicine reminder chart
  Arms: Patient-centred tailored intervention

SUMMARY:
The purpose of this study is to find out whether talking to a pharmacist on the telephone can help to support people taking medicine for a long-term condition.

DETAILED DESCRIPTION:
Non-adherence to medication is common and although some interventions have shown promise in improving adherence, the findings are inconsistent. This randomised controlled trial aims to test the effectiveness of a pharmacy-based telephone intervention compared to usual care on medication adherence and health outcomes in patients taking medicines for a long-term condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed medication(s) for at least one of the following conditions: type 2 diabetes, hyperlipidemia

Exclusion Criteria:

* Patients living outside of England
* Patients with no access to a telephone
* Patients under the age of 18
* Patients unable to give written informed consent
* Patients on drugs for dementia
* Patients showing signs of dementia or cognitive impairment in conversation
* Patients with substantial hearing or sight impairment
* Patients whose medications are ordered by a caregiver/family member
* Patients with insufficient English to take part in the telephone intervention
* Patients living with someone already taking part in the study
* Patients newly prescribed a medication for the conditions listed in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Self-reported medication adherence | 6 months

SECONDARY OUTCOMES:
Prescription refill adherence | Baseline, 6 months and 12 months
Self-reported medicine-related problems and concerns | Baseline, 3 months and 6 months
  Medicine-related problems and concerns will be assessed in a self-report questionnaire.
Beliefs about Medicines | Baseline, 3 months and 6 months
  Beliefs about medicines will be assessed in a self-report questionnaire using the Beliefs About Medicines Questionnaire (BMQ) (Horne et al. 1999).
HbA1c | Baseline and 6 months
Serum Cholesterol Levels | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nick Barber, Principal Investigator — UCL School of Pharmacy
Locations (1):
- UCL School of Pharmacy, London, United Kingdom

REFERENCES:
- [Derived] Lyons I, Barber N, Raynor DK, Wei L. The Medicines Advice Service Evaluation (MASE): a randomised controlled trial of a pharmacist-led telephone based intervention designed to improve medication adherence. BMJ Qual Saf. 2016 Oct;25(10):759-69. doi: 10.1136/bmjqs-2015-004670. Epub 2016 Jan 11. PMID 26755665